CLINICAL TRIAL: NCT06313918
Title: Exercise Therapy in Mental Disorders-study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REK nr. 428096
Record Dates: First submitted 2023-10-20; First posted 2024-03-15 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia and Related Disorders; Bipolar Disorder
Keywords: Exercise therapy; Effectiveness
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Open label, two-arm, parallel group, randomised trial, to compare standard and short HIT during 26 weeks of supervised exercise. The group will receive comprehensive follow-up to be able to carry out the 26 weeks exercise intervention program. Outcome measures will be taken at; baseline (T0), 4 weeks (T1), 12 weeks (T2), 26 weeks (T3), and 52 weeks (T4) post randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard HIT (Active Comparator): Standard 4 x 4 min HIT at treadmill. First 7 min warm-up, then 4 sessions with 4 min walking/running at 80-95% of maximal heart rate, with 3 min of active rest in between. Ending with 5 min of cooling down. Two sessions per week for 26 weeks.
  Interventions: Other: High intensity training (HIT)
- Short HIT (Experimental): Short 1 x 4 min HIT at treadmill. Starting with 7 min warm-up walking/running, then 1 session with 4 min walking/running at 80-95% of maximal heart rate, ending with 5 min of cooling down. Two sessions per week for 26 weeks.
  Interventions: Other: High intensity training (HIT)

INTERVENTIONS:
Other: High intensity training (HIT) — Please see information already included in the arm descriptions.

SUMMARY:
The study will compare standard high-intensity training with brief high-intensity training in people with schizophrenia-spectrum or bipolar disorder. The overall aim is to determine which of the two is superior in a long-term perspective.

DETAILED DESCRIPTION:
Background: Patients with severe mental disorders (SMD), including schizophrenia spectrum and bipolar disorders, frequently experience suboptimal treatment effectiveness resulting in disabling residual symptoms and cognitive challenges, and have elevated mortality risk amounting to 15-20 years of shortened life expectancy compared to the general population.

Cardiovascular disease (CVD) is a major contributor in this regard. Exercise in general improves cognitive functioning, negative symptoms, quality of life, and reduces the risk of CVD. High intensity training (HIT) has been shown to be feasible for persons with SMD, but attrition and noncompliance are substantial and likely to limit the effectiveness of HIT. A less strenuous HIT could increase adherence to the intervention, which might compensate for a slightly lower efficacy compared to standard HIT. Our study will compare standard 4x4-min HIT to a 4-min single-bout HIT session, as well as explore exercise effects on basic processes in the body. Methods: Patients with schizophrenia spectrum and bipolar disorders are eligible for participation, and those included will be randomized to 26 weeks of either 1) Standard 4 x 4 min HIT at treadmill, or 2) Short 1 x 4 min HIT at treadmill. To reduce dropout, the intervention will usually be delivered in group format, and conducted under the supervision of a physical therapist in collaboration with a postdoctor. The research group has a stable staff with research nurses, biostatisticians and researchers that will secure the dayto- day conductance of the project, including psychometric assessments, drawing of and biobanking of blood, as well as data collection and storing. Measures: Mental and cognitive symptoms, quality of life, motivation, Peak oxygen uptake (V

ELIGIBILITY:
Inclusion Criteria:

* ICD-10 schizophrenia-spectrum disorder (F2)
* ICD-10 bipolar disorder (F3)
* Capacity to provide informed consent.

Exclusion Criteria:

* Contra-indication for exercise training and testing according to the American College of Sports Medicine specifications
* Life threatening or terminal medical conditions
* Not able to carry out intervention or test procedures
* Current pregnancy
* Mothers less than 6 months post-partum.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2026-09-26 (Estimated); Study Completion 2026-09-26 (Estimated)

PRIMARY OUTCOMES:
Adherence | 26 weeks
  Proportion (number and percent) of completers at 26 weeks.

SECONDARY OUTCOMES:
Change of the Simplified Negative and Positive Symptoms Interview (SNAPSI) score | 4, 12, 26 and 52 weeks from baseline
  Symptoms of psychosis
Change of the Calgary Depression Scale in Schizophrenia score | 4, 12, 26 and 52 weeks from baseline
  Symptoms of depression
Change of the Clinical Global Impression (CGI) score | 4, 12, 26 and 52 weeks from baseline
  Overall clinical state
Change of the Global Assessment of Funtioning (GAF) score | 4, 12, 26 and 52 weeks from baseline
  Functioning
Change of quality of life (QOL10) score | 4, 12, 26 and 52 weeks from baseline
  Quality of life
Change of the International Physical Activity Questionaire (IPAQ) score | 4, 12, 26 and 52 weeks from baseline
  Physical activity
Change of the Brief Assessment of Cognition in Schizophrenia (BACS) score | 4, 12, 26 and 52 weeks from baseline
  Cognition
Change of the Behavioural Regulation in Exercise Questionaire (BREQ) score | 4, 12, 26 and 52 weeks from baseline
  Motivation
Change of the Difficulties in Emotion Regulation (DERS) score | 4, 12, 26 and 52 weeks from baseline
  Emotion regulation
Change in heart rate (beats per minute) | 4, 12, 26 and 52 weeks from baseline
  Heart rate variability
Change of maximal oxygene extraction (VO2max) | 4, 12, 26 and 52 weeks from baseline
  Aerobic capacity
Change of level of inflammatory markers in blood | 4, 12, 26 and 52 weeks from baseline
  Inflammation
Change of body weight (kilograms) | 4, 12, 26 and 52 weeks from baseline
  Body weight change
Change of hip- and waist circumference (centimetres) | 4, 12, 26 and 52 weeks from baseline
  Change of hip- and waist circumference
Change of serum glucose (mmol/L) | 4, 12, 26 and 52 weeks from baseline
  Change of serum glucose
Change of serum cholesterols (mmol/L) | 4, 12, 26 and 52 weeks from baseline
  Change of serum cholesterols
Change of serum triglyceride (mmol/L) | 4, 12, 26 and 52 weeks from baseline
  Change of serum triglyceride (mmol/L)
Change of gene expression | 4, 12, 26 and 52 weeks from baseline
  RNA
Change of methylation of DNA | 4, 12, 26 and 52 weeks from baseline
  Epigenetic changes
Change of the Young Mania Rating Scale (YMRS) score | 4, 12, 26 and 52 weeks from baseline
  Symptoms of mania

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No